CLINICAL TRIAL: NCT03844906
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study of Multiple Doses of SAGE-718 Using Ketamine Challenge to Evaluate the Electrophysiology, Safety, Tolerability, and Pharmacokinetics in Healthy Subjects
Brief Title: A Study to Assess Electrophysiology, Safety, Tolerability, and Pharmacokinetics of Multiple Doses of SAGE-718 Using Ketamine Challenge in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 718-EXM-103
Record Dates: First submitted 2018-12-19; First posted 2019-02-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAGE-718 (Experimental)
  Interventions: Drug: SAGE-718
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAGE-718 — SAGE-718 in combination with Ketamine
  Arms: SAGE-718
Drug: Placebo — Placebo in combination with Ketamine
  Arms: Placebo

SUMMARY:
This study is a Phase 1, randomized, double-blind, placebo-controlled study of multiple doses of SAGE-718 using ketamine challenge to evaluate the electrophysiology, safety, tolerability, and pharmacokinetics in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a body weight ≥50 kg and body mass index (BMI) ≥18.0 and ≤30.0 kg/m2 at screening.
2. Subject is healthy with no history or evidence of clinically relevant medical disorders as determined by the Investigator.

Exclusion Criteria:

1. Subject has any clinically significant abnormal value for hematology, clinical chemistry, or urinalysis at screening or admission.
2. Subject has a history or presence of a neurologic disease or condition, including but not limited to epilepsy, closed head trauma with clinically significant sequelae, or a prior seizure.
3. Subject has a positive screening test for alcohol or drugs of abuse (including marijuana) at screening or admission.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Changes in Electrophysiological Parameters Pre- and Post-ketamine Infusion in Participants Receiving SAGE-718 vs Placebo | From Day 1 through Day 11
Number of Participants With Changes in Auditory-Evoked Potentials Pre- and Post-ketamine Infusion in Participants Receiving SAGE-718 vs Placebo | From Day 1 through Day 11

SECONDARY OUTCOMES:
Number of Participants with the Incidence of Adverse Events and Serious Adverse Events. | Between Baseline and Day 26

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sage Investigational Site, Long Beach, California
  - Sage Investigational Site, Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.